CLINICAL TRIAL: NCT04450654
Title: Monotherapy IVIG Gamunex-C for HMG-CoA Reductase Auto-Antibody Positive Necrotizing Myopathy Treatment (The MIGHT Trial)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: University of Washington (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Principal Investigator, James S. Andrews, Assistant Professor, School of Medicine: Rheumatology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00009143
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Immune-Mediated Necrotizing Myopathy
Keywords: HMG-CoA Reductase Auto-Antibody Necrotizing Myopathy
MeSH Terms: interventions — Hizentra; Immunoglobulins, Intravenous; Albumins

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded, placebo-controlled phase 2 trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gamunex-C IVIG (Experimental): Gamunex-C IVIG dosed at 2g/kg will be given on week 0 and week 4.
  Interventions: Drug: Gamunex-C
- Placebo (Placebo Comparator): Albumin in a 1% solution at an equivalent volume to the corresponding Gamunex-C IVIG dose will be given at week 0 and week 4.
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: Gamunex-C — Gamunex-C IVIG will be given at week 0 and week 4
  Other Names: IVIG
  Arms: Gamunex-C IVIG
Drug: Albumin — 1% albumin solution dosed at equivalent volume to the corresponding weight-based Gamunex-C IVIG dose will be given at week 0 and week 4
  Arms: Placebo

SUMMARY:
This is a phase 2, pilot, randomized, placebo-controlled trial of Gamunex-C IVIG as mono-therapy for HMGCoA reductase auto-antibody positive (HMGCR) necrotizing myopathy. The trial will test the feasibility and initial efficacy of Gamunex-C IVIG mono-therapy in HMGCR necrotizing myopathy.

DETAILED DESCRIPTION:
This is a phase 2, double-blinded, randomized, placebo-controlled, multi-center trial of Gamunex-C IVIG as mono-therapy for HMGCR necrotizing myopathy. Up to 10 treatment-naïve patients will be enrolled and randomized to receive either Gamunex-C IVIG dosed at 2g/kg or placebo at week 0 and week 4. The primary efficacy outcome is the percentage of patients at week 8 with at least minimal improvement per the 2016 ACR/EULAR myositis clinical response criteria.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following inclusion criteria at screening to be eligible for participation in this study:

* Anti-HMGCR positive. Patients will be screened by commercially-available ELISA.
* Age ≥ 18 years
* Demonstrable proximal muscle weakness: score of <135 on the Proximal Manual Muscle Strength Testing 8-Muscle Group Assessment (MMT-8) (range 0-160).
* Serum creatinine kinase (CK) more than 5 times the upper limit of normal
* Muscle biopsy will not be required for eligibility in order to minimize the time to enrollment and initiation of treatment. Muscle biopsy will be obtained whenever possible as part of the standard of care.
* Subjects must be willing and able to provide written informed consent.

Exclusion Criteria:

A subject meeting any of the following exclusion criteria at screening is NOT eligible for participation in this study:

* Disease duration greater than 36 months.
* Participants taking oral or intravenous glucocorticoids where the dose has changed within 4 weeks of screening.
* Exposure to immunoglobulin treatment (IV, IM, or SubQ) in the prior 3 months
* Exposure to plasma exchange (PEX) in the prior 3 months
* Exposure to other immunosuppressive medications (e.g. methotrexate, leflunomide, azathioprine, mycophenolate mofetil) in the prior 6 months
* Exposure to rituximab or any monoclonal antibody in the prior 12 months
* Currently taking a statin medication
* History of dermatomyositis rash (either biopsy-proven, or history of photosensitive rash).
* Presence of respiratory or swallowing dysfunction due to HMGCR myopathy
* Inadequate venous access
* History of anaphylactic reactions or severe reactions to any blood-derived product
* History of intolerance to any component of the IP
* History of thrombotic complication to polyclonal IVIG therapy
* History of pulmonary embolism or deep venous thromboembolism
* History of hyperviscosity or hypercoagulable state
* History of myocardial infarction or stroke in the last 12 months
* Currently receiving anti-coagulation therapy (vitamin K antagonists, non-vitamin K oral anticoagulants [e.g. dabigatran, rivaroxaban, apixaban], parenteral anticoagulants [e.g fondaparinux]. Note that oral anti-platelet agents are allowed (e.g. aspirin, clopidogrel, ticodipine).
* Females of child-bearing potential who are pregnant, have a positive serum pregnancy test (human chorionic gonadotropin [HCG]-based assay), breastfeeding, or are unwilling to practice a highly effective method of contraception (oral, injectable or implanted hormonal methods of contraception, placement of an intrauterine device or intrauterine system, condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or true abstinence*) throughout the study.

  * True abstinence: When this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods], declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception.)
* Renal impairment (i.e., estimated glomerular filtration rate (eGFR) below 60ml/min)
* History of chronic liver disease
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels exceeding more than 2.5 times the ULN for the expected normal range for the testing laboratory, not due to HMGCR myopathy.
* Hemoglobin level <9 g/dL
* Known Immunoglobulin A (IgA) deficiency and anti-IgA serum antibodies
* History of chronic alcoholism or illicit drug abuse (addiction) in the prior 12 months
* Active psychiatric illness that interferes with compliance or communication with healthcare personnel
* Currently receiving, or having received, within 1 month prior any investigational medicinal product or device. In the case of an investigational medicinal product trial, at least five half- lives (if known) must have elapsed prior to Screening.
* Any medical condition which makes the clinical trial participation unadvisable or which is likely to interfere with the evaluation of the study treatment and/or the satisfactory conduct of the clinical trial according to the investigator's judgment. Any factor that in the opinion of the investigator would compromise the ability of the subject to complete the trial
* Weight > 120kg. Individuals weighing >100kg and ≤120kg will be eligible at the discretion of the investigators.
* History of angina pectoris or transient ischemic attack (TIA) in the last 12 months
* Wells Criteria Score for DVT of 2 or more at the time of screening.
* Wells Criteria Score for PE of 4 or more at the time of screening.
* Presence of a central, in-dwelling catheter (such as a PICC line) at the time of informed consent.
* Currently taking a nephrotoxic drug (eg gentamicin or vancomycin) at the time of informed consent.
* Severe cardiac failure at the time of informed consent.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
ACR/EULAR 2016 Clinical Response Criteria for Myositis | week 8
  The percentage of patients in each arm with at least a minimal response

SECONDARY OUTCOMES:
Manual Muscle Strength Testing (MMT-8) score | week 8
  Manual muscle strength testing in 8 muscle groups will be scored. Range 0-160, with higher scores reflecting increased muscle strength.
ACR/EULAR Clinical Response Criteria for Myositis Total Improvement Score | week 8
  The total improvement score based on ACR/EULAR 2016 criteria will be calculated. Range 0-100, with higher scores reflecting greater improvement.
HMG-CoA Reductase Auto-antibody titer level | week 8
  Autoantibody titer level will be assessed
Creatine kinase | week 8
  Serum creatine kinase level will be measured
Number of patients screened to achieve planned enrollment | 2 years
Number of days needed to enroll planned sample | 2 years
Percentage of enrolled patients completing all primary and secondary measures | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James S Andrews, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States